CLINICAL TRIAL: NCT05146323
Title: Personalization of 99mTc-Sestamibi Activities in SPECT/CT Myocardial Perfusion Imaging With the Cardiofocal SmartZoom® Collimator
Brief Title: Optimization of 99mTc-Sestamibi Activities in SPECT/CT Myocardial Perfusion Imaging
Acronym: OSPECT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-06Obs-CHRMT
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Coronary Heart Disease
Keywords: Myocardial SPECT; Sestamibi; SmartZoom; Cardiofocal collimator; Dose optimization
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This work suggests a methodology to adapt the injected radionuclide activity to the level of attenuation of each patient. The investigators propose a dose reduction adapted to the patient's weight, with no significant degradation of the image quality, in order to improve patients and staff radioprotection, standardize the image quality for easier clinical interpretation, and lead to radiopharmaceutical saving in the context of myocardial perfusion Imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent stress-test 99 mTc-Sestamibi SPECT/CT myocardial perfusion Imaging on a Siemens Intevo Bold Anger camera with the cardiofocal SmartZoom® collimator

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with myocardial perfusion Imaging in the context of coronary heart disease
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Number of counts | Day 1
  Number of counts in the myocardial region of interest

SECONDARY OUTCOMES:
Clinical evaluation | Day 1
  Medical evaluation of image quality, in order to establish a correlation between the myocardial signal level and the clinical image quality

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, Moselle, France